CLINICAL TRIAL: NCT05841433
Title: Relationship Between Blood Groups , Iron Deficiency Anemia and Helicobacter Pylori in Children.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliaa Abdelhak Shehab, Resident doctor at asset university, Assiut University
Other Study IDs: 357357
Record Dates: First submitted 2023-01-25; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Relationship Between Blood Groups , Iron Deficiency Anemia and Helicobacter Pylori in Children
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional

SUMMARY:
Iron-deﬁciency anemia (IDA) represents a global public health problem which has a signiﬁcant impact on human health and social and economic development. Inadequate iron intake, chronic blood loss and impaired iron absorption are among the causes of IDA There are an association between H. pylori infection and IDA, but the biological explanation for H. pylori infection causing iron-deﬁciency anemia remains unknown. Initially, sideropenic anemia was considered to be caused by occult blood loss due to chronic superﬁcial active gastritis caused by H. pylori, but subsequent studies did not conﬁrm this theory . H. pylori infection can cause disorders in iron assimilation and increased iron requirements. Hypoacidity caused by pangastritis and a low level of ascorbic acid in the stomach of patients infected with H. pylori may affect the absorption of iron in the duodenum . In addition, levels of lactoferrin gastric mucosa (an iron-binding protein) are high in patients infected with iron-deﬁcient H. pylori, showing a possible role between increased lactoferrin sequestration and iron utilization by the body . H. pylori also competes with the host for available food grade iron. H. pylori has several iron acquisition systems, which can capture iron available in the microenvironment of the stomach lumen . Moreover, there are studies that indicate that an iron-deﬁciency anemia which does not respond to iron therapy can be resolved by eradicating H. pylori from the stomach . ABO blood group seem to be looked into as risks for H. pylori related stomach malignancy, nevertheless, there are actually inconsistent scientific studies because of numerous confounding outcomes. Blood group antigens have the receptor properties for toxins, parasitic organisms and bacteria, exactly where this bacteria could assist in annexation or intrusion and avert multitude approval components .

DETAILED DESCRIPTION:
Iron-deﬁciency anemia (IDA) represents a global public health problem which has a signiﬁcant impact on human health and social and economic development. Inadequate iron intake, chronic blood loss and impaired iron absorption are among the causes of IDA There are an association between H. pylori infection and IDA, but the biological explanation for H. pylori infection causing iron-deﬁciency anemia remains unknown. Initially, sideropenic anemia was considered to be caused by occult blood loss due to chronic superﬁcial active gastritis caused by H. pylori, but subsequent studies did not conﬁrm this theory . H. pylori infection can cause disorders in iron assimilation and increased iron requirements. Hypoacidity caused by pangastritis and a low level of ascorbic acid in the stomach of patients infected with H. pylori may affect the absorption of iron in the duodenum . In addition, levels of lactoferrin gastric mucosa (an iron-binding protein) are high in patients infected with iron-deﬁcient H. pylori, showing a possible role between increased lactoferrin sequestration and iron utilization by the body . H. pylori also competes with the host for available food grade iron. H. pylori has several iron acquisition systems, which can capture iron available in the microenvironment of the stomach lumen . Moreover, there are studies that indicate that an iron-deﬁciency anemia which does not respond to iron therapy can be resolved by eradicating H. pylori from the stomach . ABO blood group seem to be looked into as risks for H. pylori related stomach malignancy, nevertheless, there are actually inconsistent scientific studies because of numerous confounding outcomes. Blood group antigens have the receptor properties for toxins, parasitic organisms and bacteria, exactly where this bacteria could assist in annexation or intrusion and avert multitude approval components .

ELIGIBILITY:
Inclusion Criteria:

* Children from both sexes their ages ranged from 4-18 years.
* Children who are diagnosed to have H. Pylori infection.

Exclusion Criteria:

* Children less than 4 years and more than 18 years.
* Children with chronic illnesses (e.g. CRF, CHF or chronic hemolytic anemias).
* Children who are receiving iron supplementation or multivitamins containing iron.

Ages: 4 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children from both sexes their ages ranged from 4-18 years diagnosed by H.pylori infection
Sampling Method: Non-Probability Sample
Enrollment: 101 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of seropositive helicopacter pylori infection and the frequencies of ABO blood groups and iron deficiency anemia in helicopacter pylori seropositive children. | baseline
  by Lohman technique , height and weight were recorded for children without shoes and wearing light clothes, standing straight, with their weight uniformly distributed on both feet and their arms hanging freely on the sides. A digital scale (model 881; Seca, Hamburg, Germany).
  Height measurements in centimeters. Body mass index (BMI) to age was obtained. Anemia was defined according to (WHO) age criteria; that is, hemoglobin level of <11 g/dL (110 g/L) in children <5 years, <11.5 g/dL (115 g/L) in children with ages between 5 and 12 years and <12 g/dL (120 g/L) for patients with ages between 12 and 18 years old. Serum ferritin level was measured using electro chemiluminescence (Elec Sys 2010 analyzer; Roche Diagnostics, Mannheim, Germany), and Serum iron level and total iron binding capacity (TIBC) were determined by CobasIntegra700 analyzer (Roche Diagnostics, Basel, Switzerland). Iron deficiency anemia (IDA) was defined as serum ferritin level of <-2SD for age.